CLINICAL TRIAL: NCT04233060
Title: A Phase I, Multi-center, Open-label, Dose Escalation Study of CS3005 in Subjects With Advanced Solid Tumors
Brief Title: A Study of CS3005 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3005-101
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS3005 (Experimental)
  Interventions: Drug: CS3005

INTERVENTIONS:
Drug: CS3005 — CS3005 will be orally administrated twice daily (BID) until PD, unacceptable toxicity, withdrawal of informed consent, or until maximum treatment duration per protocol (2 years)

SUMMARY:
A Phase I, Multi-center, Open-label, Dose Escalation Study of CS3005 in Subjects with Advanced Solid Tumors

ELIGIBILITY:
General

1. Be willing and able to provide written informed consent form for the trial.
2. Male or female between 18 to 75 years of age.
3. Ability to comply with requirements of the protocol, as assessed by the investigator.
4. Subjects who were histologically confirmed advanced solid tumor shall have progressed disease and/or experienced intolerance from prior standard therapies, or for whom no standard of care (SoC) therapies exist.
5. Subject must have at least one measurable lesion by CT or MRI; radiographic tumor assessment should be performed within 28 days prior to the first dose of study treatment.
6. ECOG performance status score of 0 or 1
7. Prior immunotherapy is allowed
8. Subjects who have previously received anti-tumor therapy will only be enrolled if the toxicities from the previous treatment have returned to the baseline level or NCI CTCAE v 5.0 grade ≤1.
9. Subject must have adequate organ function as indicated by the following laboratory values, G-CSF or other relevant medical support within 14 days before the administration of the investigational product
10. Subjects with active hepatitis B or active hepatitis C must receive antiviral treatment and pass the HBV DNA titer test and HCV RNA test before being enrolled. The subject should be willing to continue effective anti-viral treatment during the study.
11. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result. Either Female or male subjects must agree to use adequate contraceptive measures.

Exclusion Criteria:

1. Has disease that is suitable for local treatment administered with curative intent
2. Has a history of a second malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
3. Patients with any condition that impairs their ability to take oral medication.
4. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. Subjects with active, known, or suspected autoimmune disease in the past 3 years prior to the start of treatment.
6. History of active tuberculosis, both pulmonary and extrapulmonary.
7. Clinically Significant history of cardiac disease within 6 months prior to 1st dosing, myocardial infarction within the previous year, or current cardiac ventricular arrhythmias requiring medication.
8. Subjects with ascites, pleural effusion, pericardial effusion which cannot be reversed by appropriate interventions.
9. Subjects with any active infections requiring systemic therapy within 2 weeks prior to the initiation of the study treatment.
10. Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
11. History of organ transplant that requires the use of immunosuppressive treatment.
12. For post immunotherapy patients, with prior ≥ Grade 3, serious, or life-threatening immune-mediated reactions following prior anti-PD-(L)1 or other immune-oncology therapies.
13. Subjects who have received systemic anti-tumor treatments 21 days prior to the initiation of the study treatment.
14. Subjects who have received treatment with approved anti-tumor Chinese herbal medicine or Chinese prepared.
15. Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications.
16. Has received treatment with non-selective adenosine antagonist or A2a receptor antagonist.
17. Concurrent administration of strong inhibitors or inducers of CYP3A4 and CYP1A2 is not permitted

For more information regarding trial participation, please contact at cstonera@cstonepharma.com

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of first dose to 30 days (±7 days) after last dose of CS3005, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, PhD, Study Director — CStone Pharmaceuticals
Locations (1):
- Scientia Clinical Research Ltd, Sydney, New South Wales, Australia